CLINICAL TRIAL: NCT00423267
Title: A Multicenter, Randomized, Controlled, Double-Blind, Double-Dummy, Two-Arm Study of Posaconazole vs Fluconazole in the Treatment of Coccidioidomycosis
Brief Title: POS vs FLU for First Line Treatment of Coccidioidomycosis (Study P04558Am1)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04558
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2010-06-30 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Coccidioidomycosis
MeSH Terms: conditions — Coccidioidomycosis | interventions — posaconazole; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Posaconazole (Experimental): Eligible subjects will be stratified at Baseline by disease site (skeletal, lung, or soft tissue) and by immune status (immunocompromised or non-immunocompromised) and will then be randomly assigned to receive Posaconazole 400 mg orally (PO) (oral suspension 40 mg/mL) administered twice daily with meals or oral nutritional supplements for 12 months.
  Interventions: Drug: Posaconazole
- Fluconazole (Active Comparator): Eligible subjects will be stratified at Baseline by disease site (skeletal, lung, or soft tissue) and by immune status (immunocompromised or non-immunocompromised) and will then be randomly assigned to receive Fluconazole 400 mg PO (given as two 200-mg oral encapsulated tablets) administered once daily for 12 months. Fluconazole treatment or placebo only occurred during Period A.
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole 400 mg orally (PO) (oral suspension 40 mg/mL) administered twice daily with meals or oral nutritional supplements for 12 months
  Arms: Posaconazole
Drug: Fluconazole — Fluconazole 400 mg PO (given as two 200-mg oral encapsulated tablets) administered once daily for 12 months
  Arms: Fluconazole

SUMMARY:
To evaluate the safety of posaconazole (POS) in the treatment of coccidioidomycosis. Period A consisted of 2 blinded arms, posaconazole and fluconazole. Recruitment was stopped, and participants in Period A may have been eligible to roll over to an open-label, non-comparitive Period B. During Period B, participants received posaconazole for a treatment duration not to exceed 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Thirteen years of age or older, 34 kg (75 lb) or more, either sex, and any race;
* Coccidioides immitis (C. immitis) or Coccidioides posadasii (C. posadasii) identified by culture or microscopic examination from skeletal disease, chronic active pulmonary disease, or soft tissue disease;
* Coccidioidomycosis score of >=6;
* Clinical laboratory safety tests within normal limits or clinically acceptable to the sponsor;
* Free of any clinically significant disease that would interfere with study evaluations;
* Willing to give written informed consent and able to adhere to study medication dose, mandatory procedures (including human immunodeficiency virus (HIV) testing), and visit schedules;
* Able to swallow food or a nutritional supplement;
* Use of a medically accepted method of contraception;
* Negative serum pregnancy test at Screening and negative urine pregnancy test at Randomization;
* Women of childbearing potential not currently sexually active must agree to use a medically accepted method of contraception should they become sexually active while participating in the study.

Exclusion Criteria:

* Key Exclusion Criteria

Excluded Medications at Enrollment

* Medications that are known to interact with POS or FLU and that may lead to serious or life threatening side effects within 7 days prior to initiating study drug;
* Medications known to lower the serum concentration/efficacy of azole antifungals within 7 days prior to study drug start;
* Prior investigational drug use or biologic product administration within 30 days before study drug start;
* Prior antifungal treatment for the current episode of infection with a total cumulative dose of >=8 g of any azole, >=4 mg/kg of amphotericin B deoxycholate, or >=20 mg/kg of lipid amphotericin B;
* Antiretrovirals that are substrates of CYP3A4 administered to HIV-positive subjects, as it is not currently known how POS or FLU may affect such drugs or the potential to cause adverse reactions.

  * Excluded Concomitant Conditions
* Immediately life-threatening coccidioidomycosis;
* Confirmed or suspected meningeal coccidioidomycosis;
* Pulmonary coccidioidomycosis in HIV-negative subjects for less than 3 months;
* Any condition requiring use of prohibited drugs;
* Cluster of Differentiation 4 (CD4) count of <200 cells/mm3 or any auto-immune deficiency syndrome (AIDS)-defining illness in HIV-positive subjects in the prior 30 days.

  * Excluded Baseline Laboratory Studies
* Moderate or severe liver dysfunction (aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times upper limit of normal (ULN)) or a total bilirubin level or direct bilirubin > 3 times ULN plus ALT or AST >2 times ULN (Hy's Rule);
* Moderate or severe renal dysfunction (creatinine clearance (CrCl) <20 mL/min) or dialysis required or expected to be required within the study period;
* Electrocardiogram (ECG) with a prolonged QTc interval by manual reading: QTc >450 msec for males and QTc >470 msec for females.

  * General Exclusion Criteria
* Prior enrollment in this study or other POS studies;
* Failed treatment with FLU or POS at any time in the past;
* History of hypersensitivity or idiosyncratic reactions to azole drug therapy;
* Women who are pregnant, intend to become pregnant, or are breast-feeding;
* Situation or condition that may interfere with optimal participation in the study;

Part of the staff personnel directly involved with this study;

* Family member of the investigational study staff.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Posaconazole: Eligible subjects will be stratified at Baseline by disease site (skeletal, lung, or soft tissue) and by immune status (immunocompromised or non-immunocompromised) and will then be randomly assigned to receive Posaconazole 400 mg orally (PO) (oral suspension 40 mg/mL) administered twice daily with meals or oral nutritional supplements for 12 months. One subject from period A declined to participate in the amended protocol and discontinued study treatment after 12 months of study drug administration.
- Fluconazole: Eligible subjects will be stratified at Baseline by disease site (skeletal, lung, or soft tissue) and by immune status (immunocompromised or non-immunocompromised) and will then be randomly assigned to receive Fluconazole 400 mg PO (given as two 200-mg oral encapsulated tablets) administered once daily for 12 months. Fluconazole treatment or placebo only occurred during Period A. Participants in this arm were given posaconazole in Period B.
Period: Period A
Arm/Group | Posaconazole | Fluconazole
Started | 9 | 7
Completed | 7 | 6
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance with protocol | 1 | 0
Not completed — Administrative | 1 | 0
Period: Period B
Arm/Group | Posaconazole | Fluconazole
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Posaconazole | Fluconazole | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Treatment-emergent Adverse Events (TRAEs) That Occurred With Posaconazole (POS) or Fluconazole (FLU) in Period A
Description: Treatment-emergent adverse events are defined as new events that occur following subject entry into the study or events that worsen following study entry state.
  Treatment-related adverse events are defined as new events that occur following subject entry into the study or events that worsen following study entry state and are judged by the investigator to be possibly, probably or definitely related to study medication.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 9 | 7
Participants | 5 | 3

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)That Occurred With POS or FLU in Period A
Description: Treatment-emergent adverse events are defined as new events that occur following subject entry into the study or events that worsen following study entry state.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 9 | 7
Participants | 8 | 5

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) That Occurred With POS in Period B
Description: as for outcome 2
Time Frame: 12 months
Measure: Number; unit: Participants
Groups:
- Posaconazole: Eligible subjects will be stratified at Baseline by disease site (skeletal, lung, or soft tissue) and by immune status (immunocompromised or non-immunocompromised) and will then be randomly assigned to receive Posaconazole 400 mg PO (oral suspension 40 mg/mL) administered twice daily with meals or oral nutritional supplements for 12 months.
Arm/Group | Posaconazole
Number analyzed (Participants) | 12
Participants | 8

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (at Least a 1 Grade Shift From Baseline) That Occurred With POS or FLU in Period A
Description: Severity grading was based on Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. This is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE; Grade 2 Moderate AE; Grade 3 Severe AE; Grade 4 Life-threatening or disabling AE; Grade 5 Death related to AE.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 9 | 7
Participants
  Hematology | 4 | 1
  Liver function tests | 4 | 3
  Renal function tests | 0 | 1
  Electrolytes | 0 | 2

5. Primary Outcome: Number of Participants With Treatment-related Treatment-emergent Adverse Events (TRAEs) That Occurred With Posaconazole (POS) in Period B
Description: as for outcome 1
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 12
Participants | 3

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities (at Least a 1 Grade Shift From Baseline) That Occurred With POS in Period B
Description: as for outcome 4
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 12
Participants
  Hematology | 2
  Liver function tests | 11
  Renal function tests | 1
  Electrolytes | 0

7. Secondary Outcome: Number of Participant Discontinuations Due to Adverse Events and/or Laboratory Evaluations of Safety in Period A
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole | Fluconazole
Number analyzed (Participants) | 9 | 7
Participants | 0 | 0

8. Secondary Outcome: Number of Participant Discontinuations Due to Adverse Events and/or Laboratory Evaluations of Safety in Period B
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Arm/Group | Posaconazole Period A | Fluconazole Period A | Posaconazole Period B
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 1/12
Other Adverse Events (participants affected / at risk) | 8/9 | 5/7 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole Period A (N=9) | Fluconazole Period A (N=7) | Posaconazole Period B (N=12)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole Period A (N=9) | Fluconazole Period A (N=7) | Posaconazole Period B (N=12)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (7) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LIP DRY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (2) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0)
SWELLING (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
BRONCHITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INCISION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PAROTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VENOMOUS STING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE FATIGUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
PANIC ATTACK (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
SWELLING FACE (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
BLEEDING VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or present any interim results

of the study without the Sponsor's prior written consent. The investigator further agrees to provide review copies to the Sponsor 45 days prior to submission for publication or presentation. The sponsor has the right to review and comment. If the parties disagree concerning the appropriateness of the data analysis and presentation, and/or confidentiality, investigator agrees to meet with the sponsor to discuss and resolve.